CLINICAL TRIAL: NCT00829673
Title: A Randomized, Two-Way, Single-Dose, Open-Label Study to Evaluate the Bioequivalence of a Test Tablet Formulation of Dexmethylphenidate Hydrochloride, (10 mg), Compared to an Equivalent Dose of a Commercially Available Reference Product (Focalin®, Novartis Pharmaceuticals Corporation) in 24 Fed, Healthy, Adult Subjects
Brief Title: Dexmethylphenidate Hydrochloride Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 04163
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Dexmethylphenidate Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Dexmethylphenidate Hydrochloride
- 2 (Active Comparator): Focalin®
  Interventions: Drug: Dexmethylphenidate Hydrochloride

INTERVENTIONS:
Drug: Dexmethylphenidate Hydrochloride — 10 mg Tablet
  Arms: 1
Drug: Dexmethylphenidate Hydrochloride — 10 mg Tablet
  Other Names: Focalin®
  Arms: 2

SUMMARY:
The objective of this randomized, single-dose, two-way evaluation is to compare the bioequivalence of a test dexmethylphenidate hydrochloride formulation to an equivalent oral dose of the commercially available dexmethylphenidate hydrochloride (Focalin®, Novartis Pharmaceuticals Corporation) in a test population of 24 adult subjects under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

1. Sex: Male and Female; similar proportion of each preferred.
2. Age: At least 18 years.
3. Weight: BMI (Body Mass Index) less than or equal to 30.
4. Qualifying subjects must be in good health and physical condition as determined by medical history, complete physical examination, and laboratory tests, all obtained within four (4) weeks prior to study start. The subjects may not have a history of significant past illness expected to affect the investigation. The normal status of subjects will be confirmed by the following procedures:

   * Laboratory Tests: Hemoglobin, hematocrit, RBC, WBC, differential count, serum electrolytes (Na, K, Cl), fasting blood glucose, BUN, bilirubin,m creatinine, AST, ALT, LD, alkaline phosphatase and urinalysis. HIV, Hepatitis B, Hepatitis C, breath alcohol test, and drugs of abuse testing will be done for screening purposes only. Urine drugs of abuse testing and breath alcohol testing will be repeated at each check-in. Female subjects will have a serum pregnancy test done at screening and a urine pregnancy test prior to each study period at check-in.

   Laboratory values which are greater than ±20% of the normal range will not qualify unless specifically accepted (with comment) by the Principal Investigator. Results of HIV, Hepatitis B, Hepatitis C, and drugs of abuse must be negative or non-reactive for the subject to qualify for the study.
   * Electrocardiogram: A 12-lead electrocardiogram (ECG) will be obtained for all subjects. The original tracings, plus interpretation, will be included in the case report form packet.
5. Subjects must read and sign the Consent Form.

Exclusion Criteria

1. Subjects not complying with the above inclusion criteria must be excluded from the study.
2. In addition, any one of the conditions listed below will exclude a subject from the study:

   * History of treatment for alcoholism, substance abuse, or drug abuse within past 24 months.
   * History of malignancy, stroke, diabetes, cardiac, renal or liver disease, or other serious illness.
   * History of GERD (gastroesophageal reflux disease), stricture of the esophagus, achalasia, malabsorption syndrome, colon cancer, or chronic colitis, including Crohn's disease.
   * History of upper gastrointestinal disorder such as dysphagia, esophagitis, gastritis, ulcers.
   * History of treatment for asthma within the past five (5) years.
   * History of marked treatable anxiety, tension, agitation.
   * History of glaucoma
   * History of motor tics
   * Family history or diagnosis of tourettes syndrome
   * History of treatment with monoamine oxidase inhibitors
   * History of seizures
   * Inability to sit upright for a period of at least 30 minutes
   * Females who are pregnant or lactating
   * History of hypersensitivity to dexmethylphenidate hydrochloride, methylphenidate or any central nervous system stimulant
3. Conditions upon screening which might contraindicate or require that caution be used in the administration of dexmethylphenidate hydrochloride, including:

   * Sitting systolic blood pressure below 90 mm Hg, or diastolic pressure below 50 mm Hg.
   * Heart rate less than 50 beats per minute after a 5-minute rest in a seated position.
4. Inability to read and/or sign the consent form.
5. Treatment with any other investigational drug during the four (4) weeks prior to the initial dosing for this study.
6. Subjects who have donated blood within four (4) weeks prior to the initial dosing for this study.
7. Subjects who smoke or use tobacco products or are currently using nicotine products (patches, gums, etc.). Three (3) months abstinence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Plisco, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmethylphenidate HCl First: 10 mg Dexmethylphenidate Hydrochloride Tablets test product dosed in first period followed by 10 mg Focalin® Tablets reference product dosed in the second period.
- Focalin® First: 10 mg Focalin® Tablets reference product dosed in first period followed by 10 mg Dexmethylphenidate Hydrochloride Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Dexmethylphenidate HCl First | Focalin® First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Dexmethylphenidate HCl First | Focalin® First
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Dexmethylphenidate HCl First | Focalin® First
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmethylphenidate HCl First | Focalin® First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 11 | 7 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 2 | 6 | 8
  White | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 16 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Dexmethylphenidate HCl: 10 mg Dexmethylphenidate Hydrochloride Tablets test product dosed in either period.
- Focalin®: 10 mg Focalin® Tablets reference product dosed in either period.
Arm/Group | Dexmethylphenidate HCl | Focalin®
Number analyzed (Participants) | 23 | 23
pg/mL | 15668.17 (5081.48) | 14526.09 (4639.79)
Statistical Analysis 1: Comparison: Dexmethylphenidate HCl vs Focalin®; Test type: Non-Inferiority or Equivalence — The ANOVA model containing factors for sequence of products, subjects within sequence, periods, and products was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 107.82, 90% CI [100.24 to 115.98] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 16 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Dexmethylphenidate HCl | Focalin®
Number analyzed (Participants) | 23 | 23
pg*h/mL | 81531.55 (40876.96) | 79972.63 (35905.93)
Statistical Analysis 1: Comparison: Dexmethylphenidate HCl vs Focalin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.74, 90% CI [97.3 to 104.29] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 16 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Dexmethylphenidate HCl | Focalin®
Number analyzed (Participants) | 23 | 23
pg*h/mL | 86046.67 (49869.68) | 84376.75 (43435.19)
Statistical Analysis 1: Comparison: Dexmethylphenidate HCl vs Focalin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.5, 90% CI [97.09 to 104.03] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.